CLINICAL TRIAL: NCT00332787
Title: Childhood Depression: Remission and Relapse
Brief Title: Determining Optimal Continuation Treatment Duration for Depressed Children and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH039188 (NIH); R01MH039188 (NIH); DSIR CT-M
Record Dates: First submitted 2006-06-01; First posted 2006-06-02 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Depression
Keywords: Major Depressive Disorder
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Fluoxetine

INTERVENTIONS:
Drug: Fluoxetine

SUMMARY:
This study will determine the optimal length of continuation treatment with fluoxetine for children and adolescents with major depressive disorder, as well as the factors that may contribute to positive response during acute and continuation treatment.

DETAILED DESCRIPTION:
Depression is a serious medical illness that affects all ages and populations. However, it has only been within the last 10 years that sufficient attention has been devoted to researching treatments for depression in children and adolescents. Symptoms of depression in this age group vary, but some common signs include pretending to be sick, refusing to go to school, clinging to a parent, or worrying that a parent may die. Older children may sulk, get into trouble at school, act in a negative or grouchy way, or feel misunderstood. Recent studies on selective serotonin reuptake inhibitors (SSRIs), one class of antidepressant medications, have shown that SSRIs are effective in reducing depression symptoms. The optimal duration of treatment, however, has yet to be established. This study will determine the optimal length of continuation treatment with fluoxetine for children and adolescents with major depressive disorder, as well as the factors that may contribute to positive response during acute and continuation treatment.

Participants in this study will first attend three study visits over a 2-week period to determine eligibility. All eligible individuals will be treated with fluoxetine for 12 weeks. Dosages will be determined by the study physician and will be based on clinical response to treatment. Study visits will occur weekly for the first 4 weeks and biweekly for the remaining 2 months. Depression symptoms, general changes, and adverse reactions will be assessed. Participants whose symptoms have improved will be eligible to enter the discontinuation phase of the study, which will entail random assignment to either fluoxetine or placebo for an additional 24 weeks. Study visits will occur biweekly for 3 months and monthly for the remaining 3 months. Depression symptoms and medication side effects will be assessed at these visits.

ELIGIBILITY:
Inclusion Criteria:

* Currently being treated on an outpatient basis
* Currently attending school
* Diagnosis of non-psychotic major depressive disorder (MDD)
* Duration of illness is at least 4 weeks
* In good general medical health
* Normal intelligence

Exclusion Criteria:

* Lifetime history of any psychotic disorder, including psychotic depression
* Diagnosis of bipolar I or II disorder
* History of alcohol or substance abuse or dependence within 6 months of study entry
* Lifetime history of anorexia nervosa or bulimia
* Pregnant or breastfeeding
* Does not agree to use an effective form of contraception (i.e., IUD, birth control pills, or barrier devices)
* Any chronic medical illness requiring regular medication
* Currently taking medication with psychotropic effects (i.e., anticonvulsants, steroids, etc.), other than stable stimulant treatment
* A first degree relative has bipolar I disorder
* Previous adequate treatment with fluoxetine was ineffective (defined as at least 20 mg/day for 4 weeks)

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200
Dates: Start 2000-06; Study Completion 2005-10

PRIMARY OUTCOMES:
Measured throughout the study: Relapse
Time to relapse

SECONDARY OUTCOMES:
Measured at Weeks 12 and 36: Functioning
Baseline characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Graham J. Emslie, MD, Principal Investigator — UT Southwestern Medical Center at Dallas
Locations (1):
- Children's Medical Center at Dallas, Outpatient Psychiatry Clinic, Dallas, Texas, United States

REFERENCES:
- [Derived] Kennard BD, Mayes TL, Chahal Z, Nakonezny PA, Moorehead A, Emslie GJ. Predictors and Moderators of Relapse in Children and Adolescents With Major Depressive Disorder. J Clin Psychiatry. 2018 Mar/Apr;79(2):15m10330. doi: 10.4088/JCP.15m10330. PMID 29474007
- [Derived] Nakonezny PA, Hughes CW, Mayes TL, Sternweis-Yang KH, Kennard BD, Byerly MJ, Emslie GJ. A comparison of various methods of measuring antidepressant medication adherence among children and adolescents with major depressive disorder in a 12-week open trial of fluoxetine. J Child Adolesc Psychopharmacol. 2010 Oct;20(5):431-9. doi: 10.1089/cap.2009.0108. PMID 20973714
- [Derived] Tao R, Emslie G, Mayes T, Nakonezny P, Kennard B, Hughes C. Early prediction of acute antidepressant treatment response and remission in pediatric major depressive disorder. J Am Acad Child Adolesc Psychiatry. 2009 Jan;48(1):71-8. doi: 10.1097/CHI.0b013e318190043e. PMID 19057412
- [Derived] Kennard BD, Hughes JL, Stewart SM, Mayes T, Nightingale-Teresi J, Tao R, Carmody T, Emslie GJ. Maternal depressive symptoms in pediatric major depressive disorder: relationship to acute treatment outcome. J Am Acad Child Adolesc Psychiatry. 2008 Jun;47(6):694-699. doi: 10.1097/CHI.0b013e31816bfff5. PMID 18434919